CLINICAL TRIAL: NCT07046286
Title: Clinical Outcomes, Safety, and Cost-Effectiveness Analysis of Two Catheters (Xianrui and Medtronic) in Radiofrequency Ablation for Varicose Veins
Brief Title: Clinical Outcomes, Safety, and Cost-Effectiveness Analysis of Two Catheters (Xianrui Da and Medtronic) in Radiofrequency Ablation for Varicose Veins
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, Director of Vascular Surgery in ChengduUTCM, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChengduUTCM10
Record Dates: First submitted 2025-02-15; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Varicose Veins of Lower Limb; Venous Insufficiency of Leg; Vascular Disease，Peripheral
Keywords: varicose veins of the great saphenous veins; radiofrequency ablation; catheters
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: According to the randomization results, the experimental group will use the endovenous radiofrequency ablation catheter produced by Xianruida Medical Technology Holdings Co., Ltd., while the control group will use the ClosureFast™ endovenous radiofrequency ablation catheter produced by Medtronic Inc. to perform the surgery. Surgical information (surgery date, limb position, distance from the treatment starting point to the saphenofemoral junction, treatment length), device usage information (device name and specifications, set power, set temperature, radiofrequency emission time), product performance evaluation, and immediate technical success will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: Treatment of great saphenous vein varicosity using the Xianruida AcoArt Venous™ (Experimental): Experimental group: Xianruida Endovenous Radiofrequency Ablation Catheter Participants will receive endovenous radiofrequency ablation (RFA) using the Xianruida catheter. The procedure includes catheter insertion into the target vein under ultrasound guidance. Data on surgery date, limb position, treatment length, and device performance will be recorded.
  Interventions: Procedure: Compare the two brands of radiofrequency ablation catheters for the treatment of lower limb varicose veins.
- Control Group: Treatment of great saphenous vein varicosity using the Medtronic ClosureFast™ endoven (Active Comparator): Control group: Medtronic ClosureFast™ Endovenous Radiofrequency Ablation Catheter Participants will undergo RFA using the Medtronic ClosureFast™ catheter. The procedure is similar to the experimental arm, with the same temperature and withdrawal speed settings. Data collected will include surgery date, limb position, treatment length, and device performance.
  Interventions: Procedure: Compare the two brands of radiofrequency ablation catheters for the treatment of lower limb varicose veins.

INTERVENTIONS:
Procedure: Compare the two brands of radiofrequency ablation catheters for the treatment of lower limb varicose veins. — 1. Surgical Procedures: Standardized radiofrequency ablation (GSV/SSV closure) was carried out in both groups by the same team. Catheter parameters were set as 120°C and 1 cm/min withdrawal speed. The treatment segment of the great saphenous vein was required to be >1 cm from the skin before anesthesia. For calf varicose veins, treatment was done after great saphenous vein ablation.
     * Experimental Group: Utilized Xianruida's catheter with advanced features. Surgical and device - related information was recorded.
     * Control Group: Used Medtronic's catheter. Similar data were recorded as in the experimental group.
  2. Postoperative Management: Consistent for both groups.
     * Compression: Applied elastic bandage + Class II compression stockings.
     * Medication: Patients took oral anticoagulants and painkillers as needed, with usage details recorded during follow - up.

SUMMARY:
This study aims to systematically compare the clinical efficacy (venous closure rate and symptom relief rate), safety (perioperative and postoperative complications), and cost-effectiveness (direct medical costs) of domestic Xianruida radiofrequency catheter and imported Medtronic catheter in endovenous radiofrequency ablation for varicose veins through a single-center, prospective, non-inferiority randomized controlled trial.

DETAILED DESCRIPTION:
Background and Rationale：Varicose veins of the lower extremities are a common vascular disorder, affecting approximately 30% of the adult population globally. In China, the number of patients with varicose veins exceeds 120 million, with a higher prevalence in females (66.7%) and a trend towards younger age groups. Traditional treatment methods, such as saphenofemoral ligation and vein stripping, as well as sclerotherapy, are associated with significant trauma and a higher risk of complications, including nerve damage and thrombosis formation. In contrast, radiofrequency ablation (RFA) has emerged as a minimally invasive, effective, and safe treatment option, with a faster recovery time and fewer complications. RFA is now recommended as a first-line treatment in international guidelines.

Despite the advantages of RFA, its adoption in China remains low, with a penetration rate of less than 5%, compared to over 30% in European and American countries. The primary barriers to wider adoption include the high cost of imported equipment (with brands like Medtronic dominating over 90% of the market) and insufficient technical dissemination in grassroots hospitals. In 2022, Xianruida's venous endovenous radiofrequency ablation system was approved for market, marking the first domestic radiofrequency catheter system with independent intellectual property rights. This system features advanced technologies such as an adaptive PID temperature control algorithm, dual-system monitoring, and optimized heating curves, enabling faster heating times (20% shorter than imported devices) and more stable temperature control (fluctuation range of ±1℃), thereby reducing the risk of thermal injury.

Study Objective：The primary objective of this study is to systematically compare the clinical efficacy, safety, and cost-effectiveness of domestic Xianruida radiofrequency catheters and imported Medtronic catheters in the treatment of varicose veins using a single-center, prospective, non-inferiority randomized controlled trial (RCT). Specifically, we aim to verify whether the domestic catheter is non-inferior to the imported product in terms of therapeutic effect and whether it offers significant economic advantages. This will provide comprehensive and scientific evidence for clinical decision-making, optimize treatment strategies for varicose veins, enhance the utilization efficiency of medical resources, and improve patient outcomes.

Study Design and Methodology This study is designed as a single-center, prospective, non-inferiority, randomized controlled trial（RCT）, following the CONSORT statement. The non-inferiority margin for the primary endpoint (venous closure rate at 12 months postoperatively) is set at Δ≤10%, based on international guidelines and similar studies.

Sample Size and Calculation: The sample size is estimated based on the literature and clinical practice. Assuming a postoperative venous closure rate of 95% in the control group (Medtronic catheter), and expecting similar closure rates in the experimental group (Xianruida catheter), with a non-inferiority margin of 10%, a significance level (α) of 0.05 (two-sided), and a power (1-β) of 0.8, the required sample size is 92 patients per group. Considering a 20% dropout rate, a total of 200 patients (100 in each group) will be recruited.

Randomization and Blinding: Patients will be randomly assigned to either the experimental group (Xianruida catheter) or the control group (Medtronic catheter) using a computer-generated block random sequence (block size=4) with central randomization by an independent third party. The study will employ assessor-blinding (ultrasound physicians and follow-up nurses) and patient-blinding. Due to the nature of the procedure and differences in catheter appearance, surgeons will not be blinded, but standardized surgical procedures and training will minimize bias.

Intervention and Postoperative Management： Surgical Procedure: Both groups will undergo standardized RFA (great saphenous vein/small saphenous vein closure) performed by the same surgical team. Catheter parameters will be set according to the manufacturer's instructions (temperature 120℃, withdrawal speed 1cm/min).

Postoperative Management: All patients will receive uniform compression dressing (elastic bandage + Class II compression stockings), oral anticoagulant medication, and painkillers as needed based on the patient's condition.

Outcome Measures Primary Endpoint: Venous closure rate confirmed by ultrasound at 12 months postoperatively (complete closure: no blood flow signal; partial closure: blood flow signal <10cm).

Secondary Endpoints:

Clinical Effectiveness: VCSS score (venous clinical severity score), AVVQ score (venous disease quality of life score), and CIVIQ-20 quality of life scale at 3, 6, and 12 months postoperatively.

Safety: Intraoperative complications (vascular perforation, catheter failure), postoperative complications (pain VAS score, DVT, skin burns, swelling, numbness, and skin sensation abnormalities), and use of anticoagulant and pain medications.

Cost-Effectiveness: Direct medical costs (catheter cost + surgical consumables + hospitalization costs) and indirect social costs (time to resume normal life).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old.
2. Clinically diagnosed with primary lower extremity varicose veins, with CEAP grade C2 - C5, and requiring treatment of the great saphenous vein segment.
3. Doppler ultrasound confirms that the reflux time of the saphenofemoral vein valve is > 1.0 second.
4. Doppler ultrasound confirms that the diameter of the great saphenous vein in the supine position is > 3mm and < 12mm.
5. Only one limb of each patient is included in the study.
6. The patient signs the informed consent form and is willing to cooperate with the examinations and follow - ups specified in the protocol.

Exclusion Criteria:

1. Thrombosis in the great saphenous vein, or combined with deep vein thrombosis, or a history of deep vein thrombosis or pulmonary embolism.
2. Recurrent varicose veins after previous treatment.
3. Severe tortuosity of the great saphenous vein, with the expectation that the catheter cannot pass through.
4. Severe lower extremity ischemia (CLI).
5. Known allergy to drugs or device materials involved in the study.
6. History of cardiac pacemaker or defibrillator implantation.
7. Pregnant or breastfeeding women.
8. Currently participating in other drug or device studies.
9. Deemed unsuitable for endovenous treatment by the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Venous Closure Rate at 12 Months Post-operation | 12 months
  The venous closure rate confirmed by ultrasound 12 months after surgery, categorized as complete closure (no blood flow signal) or partial closure (blood flow signal < 10 cm).This classification is used to determine the difference in the effect of achieving venous occlusion between the two catheters.
  Unit of Measure: Percentage of closed veins (%)

SECONDARY OUTCOMES:
Change in Aberdeen Varicose Vein Questionnaire (AVVQ) Score from | 3, 6, and 12 months
  Change in AVVQ score (range 0-100) at 3, 6, and 12 months to assess patient-reported symptoms.Unit of Measure: Points on scale
Change in Venous Clinical Severity Score (VCSS) from Baseline | 3, 6, and 12 months
  Change in VCSS score (range 0-30) at 3, 6, and 12 months after surgery to assess symptom improvement.Unit of Measure: Points on scale
Change in CIVIQ-20 Score from Baseline | 3, 6, and 12 months
  Change in CIVIQ-20 score (range 0-100) at 3, 6, and 12 months to assess quality of life.Unit of Measure: Points on scale
Number of Intraoperative Complications | During surgery
  Number of events during surgery, such as perforation or catheter failure.Unit of Measure: Number of events
Number of Postoperative Complications within 30 Days | 12 months
  Number of adverse events (e.g., pain, DVT, skin burns) occurring within 12 months post-operation.Unit of Measure: Number of events
VAS Pain Score on Postoperative Days 1, 3, and 7 | Days 1, 3, and 7 post-operation
  Patient-reported pain intensity using a Visual Analog Scale (range 0-10), assessed on postoperative days 1, 3, and 7.Unit of Measure:VAS score (score on a scale)
Number of Days of Painkiller Use | Within 30 days post-operation
  The total number of days pain medications are used by each participant following surgery.Unit of Measure:Days
Total Direct Medical Costs per Patient | 12 months
  Total medical cost (in Chinese Yuan) associated with the procedure, including the cost of the catheter, disposable medical supplies, and hospitalization.Unit of Measure:CNY
Number of Days to Return to Normal Life | Within 12 months
  The number of days from the procedure until the participant resumes normal daily activities or work.Unit of Measure:Days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farah MH, Nayfeh T, Urtecho M, Hasan B, Amin M, Sen I, Wang Z, Prokop LJ, Lawrence PF, Gloviczki P, Murad MH. A systematic review supporting the Society for Vascular Surgery, the American Venous Forum, and the American Vein and Lymphatic Society guidelines on the management of varicose veins. J Vasc Surg Venous Lymphat Disord. 2022 Sep;10(5):1155-1171. doi: 10.1016/j.jvsv.2021.08.011. Epub 2021 Aug 24. PMID 34450355
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] Zhai Y, Lu YM, Lu W, Yang C. Radiofrequency ablation of the great saphenous vein in the treatment of varicose veins of the lower extremities. Ann Ital Chir. 2022;93:235-240. PMID 35503057
- [Background] Tang MJ, Zhou LY, Jia XJ, Wu JJ, Lou YB, Jin MJ, Zhu YF. [Randomized controlled study on the application effect of a new type of intravenous radiofrequency closed therapy system made in China and an imported system]. Zhonghua Wai Ke Za Zhi. 2024 Mar 1;62(3):223-228. doi: 10.3760/cma.j.cn112139-20231012-00167. Chinese. PMID 38291638
- See also: Xianruida's endovenous radiofrequency ablation device for the treatment of varicose veins has been approved for marketing — https://irnews.cfbond.com/detail.html?newsid=qmsyWGTZiPM%3D